CLINICAL TRIAL: NCT01830985
Title: A Phase 2/3 Open-label Extension Study to Evaluate Long-Term Safety and Efficacy With VX-509 in a Treat to Target Setting in Subjects With Rheumatoid Arthritis on Disease-Modifying Antirheumatic Drugs
Brief Title: A Phase 2/3 Open-label Extension Study to Evaluate Long-Term Safety and Efficacy With VX-509 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX12-509-104; 2012-004342-14 (EudraCT Number)
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 2-((2-(1H-pyrrolo(2,3-b)pyridin-3-yl)pyrimidin-4-yl)amino)-2-methyl-N-(2,2,2-trifluoroethyl)butanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm VX-509 (Experimental)
  Interventions: Drug: VX-509

INTERVENTIONS:
Drug: VX-509 — VX-509 dose may be increased every 8 weeks in a stepwise fashion from 100 to 150 mg and from 150 to 200 mg, as needed (determined by ongoing disease activity by CDAI)

SUMMARY:
This study is designed to evaluate the long-term safety and tolerability of VX-509 in subjects with active rheumatoid arthritis (RA) on DMARD therapy. This study will enroll subjects who completed a previous designated study with VX-509 (e.g., Study VX12-509-103).

DETAILED DESCRIPTION:
VX-509 is an oral, selective Janus kinase 3 (JAK3) inhibitor being developed by Vertex. In autoimmune diseases, JAK3 is an essential component of the immune signaling cascade. This cascade ultimately contributes to abnormal immune response that results in chronic inflammation and, in the case of rheumatoid arthritis (RA), irreversible damage to cartilage and bones. Selective inhibition of JAK3 offers a new disease modifying approach to the treatment of RA.

This study will follow a "treat to target" (T2T) paradigm. T2T strategies have been followed in non-rheumatologic fields for decades. T2T trials have been conducted for RA from the late 1990's, and have substantiated the concept that treating to a target is associated with a better outcome than standard of care treatment. This has led to recommendations by experts to use T2T strategies in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed the assigned study drug treatment phase of a previous VX-509 study (e.g., Study 103).
* Subjects must voluntarily sign and date the Study 104 informed consent document.
* Subject must be willing and able to comply with the scheduled visits, treatment plan, laboratory tests, contraceptive guidelines, and other study procedures.

Exclusion Criteria:

* Inflammatory and rheumatological disorders other than RA, where arthritis may be a prominent feature.
* History of any clinically significant illness that might, in the opinion of the investigator, confound the results of the study or pose an additional risk in administering study drug(s) to the subject
* History of tuberculosis (TB), regardless of history of antimycobacterial treatment.
* Planned surgery during the study.
* History of alcohol or drug abuse, or excessive alcohol consumption as determined by the investigator, during the previous 12 months before Day 1.
* Pregnant or nursing an infant or with a life partner who is pregnant, nursing, or planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Long-term safety and tolerability of VX-509 treatment | Baseline through 104 weeks
  Measured by clinical laboratory tests
Long-term safety and tolerability of VX-509 treatment | Baseline through 104 weeks
  Measured by adverse events (AEs)
Long-term safety and tolerability of VX-509 treatment | Baseline through 104 weeks
  Measured by electrocardiograms (ECGs)
Long-term safety and tolerability of VX-509 treatment | Baseline through 104 weeks
  Measured by vital signs

SECONDARY OUTCOMES:
Proportion of subjects who achieve CDAI LDA (≤10) or CDAI remission (≤2.8) | Baseline through 104 weeks
Proportion of subjects who achieve ≥20% (50%, 70%) improvement in disease severity according to the ACR criteria, using CRP (ACR20 CRP, ACR50 CRP, ACR70 CRP) | Baseline through 104 weeks
Change from baseline in DAS28 using CRP (4-component) (DAS28 4[CRP]) | Baseline through 104 weeks
Proportion of subjects with DAS28 4(CRP) <2.6 (DAS remission) | Baseline through 104 weeks
Proportion of subjects who achieve a moderate, good, or no response according to the EULAR response criteria from baseline | Baseline through 104 weeks
Percentage of subjects with decreased dose of DMARD and/or corticosteroid (if receiving), including the subsets with 50% withdrawal and with full withdrawal (dose = 0) | Baseline through 104 weeks
ACR hybrid scores | Baseline through 104 weeks
Proportion of subjects who achieve ACR20/50/70 with erythrocyte sedimentation rate (ESR) and DAS28 4(ESR) response from baseline | Baseline through 104 weeks
Proportion of subjects with DAS28 4(CRP) <3.2 (DAS LDA) from baseline | Baseline through 104 weeks
Proportion of subjects achieving a clinical remission (2011 ACR/EULAR criteria), including subsets achieving either the low joint count or simplified disease activity index (SDAI) score remission options (or both) from baseline | Baseline through week 104
Change from baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) | Baseline through 104 weeks
Change from baseline in health-related quality of life assessed by 36-Item Short Form (SF 36) Physical Component Summary score and Physical Function (PF) subscale | Baseline through 104 weeks

OTHER OUTCOMES:
Change in Outcome Measures in Rheumatology Clinical Trials (OMERACT) RAMRIS synovitis score, bone marrow edema (osteitis), erosion score, and joint space narrowing score by magnetic resonance imaging (MRI) in the designated hand | Baseline through week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Bloom, MD, FACR, FAAP, Study Chair — Vertex Pharmaceuticals Incorporated
Locations (22):
- United States (18):
  - Vertex Investigational Site, Upland, California
  - Vertex Investigational Site, Fort Lauderdale, Florida
  - Vertex Investigational Site, Venice, Florida
  - Vertex Investigational Site, West Palm Beach, Florida
  - Vertex Investigational Site, Canton, Georgia
  - Vertex Investigational Site, Decatur, Georgia
  - Vertex Investigational Site, Elizabethtown, Kentucky
  - Vertex Investigational Site, Fredrick, Maryland
  - Vertex Investigational Site, Lincoln, Nebraska
  - Vertex Investigational Site, Rochester, New York
  - Vertex Investigational Site, Greensboro, North Carolina
  - Vertex Investigational Site, Duncansville, Pennsylvania
  - Vertex Investigational Site, Charleston, South Carolina
  - Vertex Investigational Site, Memphis, Tennessee
  - Vertex Investigational Site, Katy, Texas
  - Vertex Investigational Site, San Antonio, Texas
  - Vertex Investigational Site, Webster, Texas
  - Vertex Investigational Site, Spokane, Washington
- Vertex Investigational Site, Tallinn, Estonia
- Vertex Investigational Site, Vilnius, Lithuania
- South Africa (2):
  - Vertex Investigational Site, Pretoria
  - Vertex Investigational Site, Stellenbosch